CLINICAL TRIAL: NCT00166075
Title: Mental Health Symptoms and Intimate Partner Violence
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Debra Houry, MD, MPH, Principal Investigator, Emory University
Other Study IDs: 0304-2003a; 5K23069375 (Other: Other)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Domestic Violence; Post-Traumatic Stress Disorder; Depression
Keywords: Suicidality; PTSD; depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Female ED patients: All eligible African American female patients were approached in the ED waiting room during study periods. Patients participated in the screening process via a computer kiosk. Questions regarding IPV and mental health symptoms were asked using validated tools
  Interventions: Procedure: Computer screen with community resource printout

INTERVENTIONS:
Procedure: Computer screen with community resource printout — Patients participated in the screening process via a computer kiosk. Questions regarding IPV and mental health symptoms were asked using validated tools

SUMMARY:
Using a touch screen computer, the researchers are screening emergency department patients for intimate partner violence and mental health issues.

DETAILED DESCRIPTION:
Using a touch screen computer, the researchers are screening emergency department patients for intimate partner violence and mental health issues. The researchers are looking to see if those who participate in a computer screen and are given referral lists as well as having the computer printout placed on the physician clipboard, will increase physician awareness and recognition as well as patient use of resources compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between the ages of 18-55 who present to the waiting room of the emergency department during study time periods

Exclusion Criteria:

* Psychotic
* Acutely intoxicated
* Too ill to participate
* Unable to read
* Not English speaking

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All eligible African American female patients were approached in the ED waiting room during study periods. Patients participated in the screening process via a computer kiosk. Questions regarding IPV and mental health symptoms were asked using validated tools.
Sampling Method: Non-Probability Sample
Enrollment: 569 (Actual)
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Increased levels of PTSD
Increased levels of suicidality
Increased levels of depression

CONTACTS AND LOCATIONS:
Overall Officials: Debra Houry, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Result] Houry D, Kemball R, Rhodes KV, Kaslow NJ. Intimate partner violence and mental health symptoms in African American female ED patients. Am J Emerg Med. 2006 Jul;24(4):444-50. doi: 10.1016/j.ajem.2005.12.026. PMID 16787803